Informed consent form(date:april2022)

Dear...

This interview will done in immunology and allergy department of Shiraz University of Medical Sciences under the title "efficacy of omalizumab in patients with recurrent nasal polyp. below Master's opinion professor hosein esmailzadeh for six months from 5<sup>th</sup> April 2022.

The purpose of this interview is help to treatment of patients with recurrent nasal polyp that is resistant to other medications. you as one The informed person will be selected and you will be interviewed and your participation is completely optional

• You can refuse to answer any questions you wish.

Name and signature of the researcher :.....

- If you leave the study, your treatment relationship with the treatment center and medical staff will not be damaged and the usual treatment methods will continue for you.
- You will not be charged for participating in this research and if you wish, you can benefit from the results at the end of the project.
- The researchers of this study will keep all information about you confidential and will use the results only for this study. The general and group results of this research will be published without mentioning my name and details.
- Participating in this research does not pose any potential risk or harm to you.
- The researcher needs your help to conduct this research and undertakes to consider the relevant ethical principles in conducting the research.

If you have any problems, objections or suggestions to those involved or the research process, you can contact the Research Ethics Committee of Shiraz University of Medical Sciences at: - Shiraz - Zand St. - next to the Red Crescent - Shiraz University of Medical Sciences Central Building - 7th floor Contact Research and Technology and present your problem orally or in writing.

This form of information and informed consent has been prepared in two copies and after signing one copy will be given to you and the other copy will be given to the executor or researcher.

Thank you for accepting to participate in this research without any expectations (financial or privilege) and whenever you have a question with the number 09171153977 Contact me.

| I In view of the above and gaining sufficient knowledge, I declare my informed and voluntary |
|---|
| consent to participate in the above research project. |
| Mobile phone (interviewee): |
| Phone: |
| Address: |
| email: |
| Signature and date: |

Date:.....